CLINICAL TRIAL: NCT03459495
Title: Investigation of the Efficacy of Therapeutic Ultrasound in the Treatment of Migraine; Prospective, Randomized, Placebo Controlled, Double-blind Study
Brief Title: Therapeutic Ultrasound in the Treatment of Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Burcu Metin Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-KAEK-2018-1/25
Record Dates: First submitted 2018-03-01; First posted 2018-03-09 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Migraine; Ultrasound
Keywords: migraine, therapeutic ultrasound, pain, disability
MeSH Terms: conditions — Migraine Disorders; Pain | interventions — Ultrasonic Therapy

STUDY DESIGN:
Intervention Model Description: prospective,randomized,placebo- controlled, double blind
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A: ultrasound group
  Interventions: Device: therapeutic ultrasound
- Group P (Placebo Comparator): Group P: placebo ultrasound group
  Interventions: Device: placebo ultrasound

INTERVENTIONS:
Device: therapeutic ultrasound — Patients in the ultrasound group will be administered to the posterior neck region for 5 minutes in pulsed mode (pulse rate 1: 1) at 1 MHz, 1.5 W / cm2. The treatment will be done 5 days a week for a total of 10 days
  Arms: Group A
Device: placebo ultrasound — When the ultrasonic device is in the closed position, the ultrasonic probe will be applied for 5 minutes in the posterior neck region of the patients. The treatment will be done 5 days a week for a total of 10 days.
  Arms: Group P

SUMMARY:
Headache affects the daily quality of life of patients. It has been reported that headaches may be associated with neck muscles, neck movements and trigger points in the neck Drug and non-drug treatments can be used today in the treatment of headaches. Various physical therapies are applied to cranial and cervical regions in non-drug therapies. Therapeutic ultrasound, Transcutaneous Electrical Nerve Stimulation (TENS), Hotpack and manipulation are some of them.This is a randomised placebo- controlled trial to determine the efficacy of the therapeutic ultrasound in the treatment of migraine.

DETAILED DESCRIPTION:
Evidence from controlled studies suggests that non-invasive physical therapies may help prevent headaches. Therapeutic ultrasound studies have generally been used in combination with other physical therapies.

Therapeutic ultrasound is known to act in two different ways, thermal and non-thermal. With thermal effect, it is possible to reduce pain and joint joints and increase local blood flow, while stimulating tissue regeneration, soft tissue repair, blood flow regulation in chronic ischemic tissues and protein synthesis with nonthermal effect. In addition, its effect on inflammation accelerated repair by affecting cell activities, altering platelet membrane permeability, leading to the release of serotonin and accelerating wound healing.

The aim of this study is to determine whether therapeutic ultrasound is superior to placebo ultrasound in the treatment of migraine.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 20-65 years
* Patients diagnosed with migraine according to the International Headache Society (IHS) criteria

Exclusion Criteria:

* Patients with bleeding disorders,
* Patients with mental disorders,
* Patients with malignancy,
* Patients with uncontrolled hypertension,
* Patients with uncontrolled diabetes mellitus,
* Patients with infection,
* Patients who underwent surgery in the posterior cranial region and cervical vertebra.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) | 4 months
  It is commonly used to measure the severity of the patients' pain. It consists of a line 10 cm. long and marked with numbers from 0 to 10. The patient is asked to mark the point corresponding to the severity of the pain on this line in the range from 0 (no pain) to 10 (most severe pain).
Migraine Disability Assessment Questionnaire Score (MIDAS) | 4 months
  The Migraine Disability Assessment (MIDAS) questionnaire is a brief, self-administered questionnaire designed to quantify headache-related disability over a 3 month period. The MIDAS score is based on five disability questions in three dimensions: questions one and two assess the number of missed or significant limitations to activity (defined as at least 50% reduced productivity) days due to headache in school or paid work activities (school/job dimension); questions three and four assess the number of missed or significant limitations to activity (defined as at least 50% reduced productivity) days due to headache in housework activities (housework dimension); question five assesses missed days due to headache in family, social, or leisure activities (social dimension).
  0 to 5 - MIDAS Grade I, Little or no disability 6 to 10 - MIDAS Grade II, Mild disability 11 to 20 - MIDAS Grade III, Moderate disability 21+ - MIDAS Grade IV, Severe disability

SECONDARY OUTCOMES:
paracetamol consumption | 4 months
the number of migraine attacks per month. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Metin Ökmen, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- Burcu Metin Ökmen, Bursa, Turkey (Türkiye)